CLINICAL TRIAL: NCT05759260
Title: Does Exercise Training Mostly Unmask Congenital Long QT Syndrome or Simply Reveals a Novel Form of Acquired Long QT Syndrome in Genetically Predisposed Youngsters Practicing Sports?
Brief Title: QT Interval in Athletes
Acronym: ERAS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 26M621
Record Dates: First submitted 2023-02-21; First posted 2023-03-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: QT Prolongation
Keywords: QT interval; Genetics; Long QT syndrome
MeSH Terms: conditions — Long QT Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Athletes with QT interval prolongation
  Interventions: Other: Observation
- Controls: Athletes without QT interval prolongation
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation

SUMMARY:
QT interval prolongation occurs in athletes and causes concerns, as it may indicate the life-threatening long QT syndrome (LQTS). Clinical and genetic testing identify those clearly affected by LQTS but in many no disease-causing mutations are found and diagnosis remains uncertain while they are barred from competitive sports. The investigators hypothesize that several cases represent an acquired form of LQTS, akin to drug-induced LQTS, caused by exercise training acting as a trigger or "second hit" on a genetic predisposition. The investigators will use next generation sequencing to screen major and minor LQTS genes plus common and rare variants modulating the QT interval in athletes with a QTc>450ms (cases) and in those with a QTc<430ms (controls). Thus, the investigators will quantify the presence of LQTS in athletes and will also focus on those who normalize their QTc after detraining, as this points to activation of stretch-receptors. The investigators will clarify QT prolongation in athletes and contribute to correct diagnosis.

DETAILED DESCRIPTION:
Background - In Italy, by law, long QT syndrome (LQTS) precludes sport participation. The Center for Cardiac Arrhythmias of Genetic Origin - Istituto Auxologico Italiano serves as referral center for sport cardiologists who certify that youngsters can practice competitive sports. Among athletes, QT interval prolongation has been frequently reported but its prevalence varies greatly from 3/1,000 to 6% based on surface ECG without genetic studies. Indeed, the presence of LQTS-causing mutations has never been quantified. Furthermore, whether this observed QT prolongation is related to training or to a latent form of LQTS has never been established. This has impacted on athlete-specific ECG criteria guidelines to distinguish between physiological or pathological values. The investigators hypothesize that QT prolongation may be an expression of "acquired" LQTS in which exercise may unmask a genetic predisposition, similar to what drugs do in drug-induced LQTS. This is supported by the investigators' observation that, following detraining, a relevant number of youngsters, all mutation-negative, normalize their QT interval. This raises the possibility that this "training-induced" QT prolongation could represent a genetic predisposition related to the activation of myocardial stretch receptors which would increase the inward calcium current and thereby prolong action potential duration. This would manifest itself as a prolongation of the QT interval on the ECG and would imply a training-induced reversible phenomenon. If recognized, this would avoid many incorrect diagnoses of LQTS.

Hypothesis and Specific Aims - Three hypotheses constitute the investigators main one, namely that QT prolongation in athletes may represent genetic variability modulated by exercise and not evidence of congenital LQTS.

The first hypothesis relates to the occurrence of prolonged QT intervals among athletes: often just a borderline prolongation but sometimes so significant to suggest LQTS. As LQTS is characterized by life-threatening arrhythmias triggered by physical or psychological stress, a correct diagnosis when dealing with youngsters practicing competitive sports is imperative. Quantification is needed and this requires genetic testing because QT prolongation in athletes cannot be automatically equated to LQTS. Among young athletes with QT prolongation the investigators expect to find both genotype-negative and genotype-positive individuals, the latter even among those with borderline QT prolongation. The results will allow to quantify the prevalence of LQTS mutation carriers (MCs) among young athletes and this early diagnosis will protect them from life-threatening arrhythmias. Sport physicians will thus be alerted to the importance of measuring the QT interval.

The investigators' second hypothesis is that, similar to drug-induced LQTS, rare or common functional variants in LQTS-associated genes may predispose to QT interval prolongation following exercise training. These variants confer either a clearly pathological (congenital) or a subclinical (exercise-induced) susceptibility. Drug-induced QT prolongation manifests itself in just a few susceptible patients receiving an IKr blocking drug. Similarly, exercise training could unmask this propensity either in "silent mutation carriers", i.e. true LQTS patients manifesting the disease only with a trigger such as exercise, or in individuals with a genetically-determined susceptibility to increase QT interval duration that needs a second-hit to manifest but which can be completely reversed once the trigger is eliminated. The third hypothesis, tightly related to the second, originates from the investigators' repeated observations of cases sharing the following features: marked QT prolongation strongly suggesting LQTS, no personal nor family history of arrhythmic events, mutation-negative, and QTc normalization after 6 or more months of detraining. The pattern is very consistent and clearly not a chance event.

Normalization following detraining suggests that prolongation was caused by training. The investigators posit that this phenomenon is due to a genetic predisposition. During exercise training the heart is exposed to substantial mechanical stress, i.e. application of forces with shear, pressure and stretch components, and responds with mechanosensitive modulation of its main regulatory processes. Mechano-sensitivity of heart rhythm, or mechano-electric feedback, is orchestrated by diverse types of stretch-activated ion channels. Among them, voltage-gated cation selective channels that normally conduct the main ionic currents determining QT duration, such as ICaL and INa. Repeated exercise is expected to initiate a mechano-electric feedback loop resulting in a reflex increase in the release of intracellular calcium which, in turn, by prolonging the plateau phase of the action potential will prolong the QT interval on the surface ECG. These effects can explain the phenomenon of transient and reversible QT prolongation which, by occurring in just a few athletes, strongly suggests a genetic predisposition. This hypothesis implies that these youngsters will no longer be labeled as "affected by LQTS"; there will be novel insights on the role of the stretch-activated channels and, a mechanistic explanation would be provided for a puzzling clinical phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Athletes
* QTc interval > 450 msec (cases) or < 430 msec (controls)

Exclusion Criteria:

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Athletes
Sampling Method: Non-Probability Sample
Enrollment: 869 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Genetic differences | At enrolment
  Quantification of MCs and non-mutation carriers (NMCs) among the young athletes with a QTc> 450 ms to define the LQTS prevalence in athletes and to identify an adequate cut-off for likely pathological QTc prolongation in athletes.

SECONDARY OUTCOMES:
Predisposition to QT prolongation | At enrolment
  Identification of genetic variants associated with predisposition to prolong the QT interval following exercise training.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano - Center for Cardiac Arrhythmias of Genetic Origin, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwartz PJ, Ackerman MJ. The long QT syndrome: a transatlantic clinical approach to diagnosis and therapy. Eur Heart J. 2013 Oct;34(40):3109-16. doi: 10.1093/eurheartj/eht089. Epub 2013 Mar 18. PMID 23509228
- [Background] Itoh H, Crotti L, Aiba T, Spazzolini C, Denjoy I, Fressart V, Hayashi K, Nakajima T, Ohno S, Makiyama T, Wu J, Hasegawa K, Mastantuono E, Dagradi F, Pedrazzini M, Yamagishi M, Berthet M, Murakami Y, Shimizu W, Guicheney P, Schwartz PJ, Horie M. The genetics underlying acquired long QT syndrome: impact for genetic screening. Eur Heart J. 2016 May 7;37(18):1456-64. doi: 10.1093/eurheartj/ehv695. Epub 2015 Dec 28. PMID 26715165
- [Background] Schwartz PJ, Woosley RL. Predicting the Unpredictable: Drug-Induced QT Prolongation and Torsades de Pointes. J Am Coll Cardiol. 2016 Apr 5;67(13):1639-1650. doi: 10.1016/j.jacc.2015.12.063. PMID 27150690
- [Background] Peyronnet R, Nerbonne JM, Kohl P. Cardiac Mechano-Gated Ion Channels and Arrhythmias. Circ Res. 2016 Jan 22;118(2):311-29. doi: 10.1161/CIRCRESAHA.115.305043. PMID 26838316